CLINICAL TRIAL: NCT02018406
Title: Establishment of Clinical Basis for Hematopoietic Growth Factors Therapy in Brain Injury
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2010-0468
Record Dates: First submitted 2013-10-30; First posted 2013-12-23 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Neurological Diseases; Ischemic Stroke; Hemorrhagic Stroke; Cerebral Palsy; Atypical Parkinson Disease
Keywords: Hematopoietic Growth Factors (EPO, G-CSF),; Neurological Diseases,; Neurorehabilitation,; Neurotrophic and Neuroprotective Effects
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Cerebral Palsy; Parkinson Disease, Familial, Type 1 | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention Group
  Interventions: Drug: Combination injection of EPO and G-CSF
- Control (Placebo Comparator): Control Group
  Interventions: Drug: Injection of normal saline

INTERVENTIONS:
Drug: Combination injection of EPO and G-CSF — Subcutaneous EPO(300 U/kg)+G-CSF(10 μg/kg) injection once a day, 5 times a cycle (a week), total 3 cycles for 3 months.
  Arms: Intervention
Drug: Injection of normal saline — Subcutaneous normal saline injection once a day, 5 times a cycle (a week), total 3 cycles for 3 months.
  Arms: Control

SUMMARY:
The purpose of our study is to determine the safety and efficacy of the combination of erythropoietin (EPO) and granulocyte-colony stimulating factors (G-CSF) in patients with neurological diseases. To be specific, our clinical study is expected that the combination injection of EPO and G-CSF shows neurotrophic and neuroprotective effects by facilitating endogenous repair process in patients with neurological diseases including stroke, cerebral palsy, or atypical parkinsonism. Therefore, we will apply our original treatment technique in patients with neurological diseases, which is expected to overcome current ethical and technical limitations of less evidenced functional recovery, hematological changes, and side effects. Eventually, We will establish a comprehensive clinical background about neurotrophic and neuroprotective effects of this hematopoietic growth factors therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old
* Voluntary participants
* Neurological diseases including stroke, cerebral palsy, or atypical parkinsonism, at least 3 months after their onset
* Participants who got previous EPO+GCSF injection at least 6 months ago.

Exclusion Criteria:

* Under 20 years old
* Participants who can not voluntarily consent
* Encephalopathy including brain tumor and infection
* Warfarin (coumadin) medications
* Leukopenia, Thrombocytopenia, Polycythemia
* Malignant diseases, Malignant hypertension, Myeloproliferative disorder, Septic embolism, Hyperkalemia
* Hepatic or Renal dysfunction, Serum creatinine>3mg/dl
* Allergic reactions against to exogenous EPO and G-CSF
* Involved in a exclusion criteria for MRI test
* A women who is pregnant or on breast feeding
* Body temperature over 38°C
* Blood pressure over 140/90 mmHg at pre-treatment
* Blood pressure over 160/100 mmHg during intervention
* Hb > 15 g/dL at pre-treatment
* Hb > 17 g/dL during intervention
* Pneumonia detected by X-ray test
* Recurrent history of aspiration pneumonia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Vital Sign | 5th day, 30th day during a cycle, and 6 months after pretest
  (1) Value of Systolic and Diastolic Blood Pressure, (2) Value of Pulse Rate, (3) Value of Respiratory Rate, (4) Value of Body Temperature.
  Vital Sign is tested to confirm the safety of the combination of EPO and G-CSF.
Hematological Test | 5th day, 30th day during a cycle, and 6 months after pretest
  (1) Value of Complete Blood Cells at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest, (2) Value of Reticulocyte at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest, (3) Value of Erythrocyte Sedimentation Rate at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest, (4) Value of C-Reactive Protein at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest, (5) Value of Electrolyte and Routine Chemistry at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest, (6) Value of Prothrombin Time and Activated Partial Thromboplastin Time at pre-treatment, 5th day, 30th day during a cycle (total three cycles), and 6 months after pretest.
  Hematological Test is tested to confirm the safety of the combination of EPO and G-CSF.
Chest and Heart Evaluation | at pre-treatment and 6 months after pretest
  (1) Chest X-ray finding at pre-treatment and 6 months after pretest, (2) Electrocardiography finding at pre-treatment and 6 months after pretest.
  Chest and Heart Evaluation is tested to confirm the safety of the combination of EPO and G-CSF.

SECONDARY OUTCOMES:
Hematological Test | 5th day, 30th day during a cycle, and 6 months after pretest
  (1) Value of Erythropoietin Level, (2) Value of CD34+ cells.
  Value of Erythropoietin Level and CD 34+ Cells are tested to demonstrate the hematological changes and effectiveness of the combination of EPO and G-CSF.
Physical Assessment | at pre-treatment, 3 months, and 6 months after pretest
  (1) Score of Muscle Strength with Manual Muscle Testing, (2) Score of Joint Mobility with Range of Motion Test, (3) Score of Muscle Spasticity with Modified Ashworth Scale.
  Physical Assessment is tested to identify functional recovery of patients by neurotrophic and neuroprotective effects of the combination of EPO and G-CSF.
Occupational Assessment | at pre-treatment, 3 months, and 6 months after pretest
  Score of Activities of Daily Living with Modified Barthel Index, Functional Independence Measure.
  Occupational Assessments is tested to identify functional recovery of patients by neurotrophic and neuroprotective effects of the combination of EPO and G-CSF.
Psychological Assessment | at pre-treatment and 6 months after pretest
  Score of Psychological Status with Mini-Mental Status Examination, Memory Quotient, Geriatric Depression Scale, if necessary
  Psychological Assessments are tested to identify functional recovery of patients by neurotrophic and neuroprotective effects of the combination of EPO and G-CSF.
Verbal Assessment | at pre-treatment and 6 months after pretest
  Score of Verbal Function with Aphasia Quotient, Boston Naming Test, Multi-dimensional Voice Performance, if necessary.
  Verbal Assessments are tested to identify functional recovery of patients by neurotrophic and neuroprotective effects of the combination of EPO and G-CSF.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Im SH, Yu JH, Park ES, Lee JE, Kim HO, Park KI, Kim GW, Park CI, Cho SR. Induction of striatal neurogenesis enhances functional recovery in an adult animal model of neonatal hypoxic-ischemic brain injury. Neuroscience. 2010 Aug 11;169(1):259-68. doi: 10.1016/j.neuroscience.2010.04.038. PMID 20610036
- [Background] Cho SR, Benraiss A, Chmielnicki E, Samdani A, Economides A, Goldman SA. Induction of neostriatal neurogenesis slows disease progression in a transgenic murine model of Huntington disease. J Clin Invest. 2007 Oct;117(10):2889-902. doi: 10.1172/JCI31778. PMID 17885687
- [Background] Seo JH, Kim H, Park ES, Lee JE, Kim DW, Kim HO, Im SH, Yu JH, Kim JY, Lee MY, Kim CH, Cho SR. Environmental enrichment synergistically improves functional recovery by transplanted adipose stem cells in chronic hypoxic-ischemic brain injury. Cell Transplant. 2013;22(9):1553-68. doi: 10.3727/096368912X662390. Epub 2013 Feb 4. PMID 23394350